CLINICAL TRIAL: NCT04694157
Title: Implication of Cardiac Shock Wave Therapy on Coronary Artery Disease Patients - An Observational Long-term Study
Brief Title: Implication of Cardiac Shock Wave Therapy on Coronary Artery Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 121-2016004-2
Record Dates: First submitted 2020-04-17; First posted 2021-01-05 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; myocardial ischemia; cardiac shock wave therapy; myocardial perfusion imaging
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum to test cardiac enzyme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: The treatment group will receive cardiac shock wave therapy. The CSWT entire treatment will period last 3 months with 9 sessions. CSWT will administered in the first week, followed by a 3-week non-treatment interval.
  Interventions: Device: cardiac shock wave therapy

INTERVENTIONS:
Device: cardiac shock wave therapy — Two target segments of left ventricle will be chosen for all participants. In each target segment, 9 sties will be administered with 200 shots at each site. Low-intensity SW (200 impulses/spot; energy flux 0.09 mJ/mm2), will be administered under electrocardiographic R-wave gating. The entire treatment period will last 3 months with 9 sessions. CSWT will be administered in the first week, followed by a 3-week non-treatment interval.

SUMMARY:
CAD is a challenging affliction which has a high annual morbidity rate in China and the world. Severe CAD may lead to compromised cardiac function, decreased exertional capacity and poor quality of life (QOL). The most common treatment for CAD is medication, percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG). However, some patients had long-term of history with complex severe artery lesions, they are not candidate for redo interventional therapy. Cardiac shock wave therapy (CSWT) is an exploring therapy used globally for CAD patients, which is known for its safety, non-invasiveness and effectiveness.The previous RCT from the investigators' team has already finished, and results are in submission processing.

This is a prospective, single arm, observational study design. CAD patients will be enrolled consecutively. The entire treatment period will last 3 months with 9 sessions. Outcomes are assessed as efficacy outcomes and safety outcomes. Efficacy outcomes include symptom (CCS score, NYHA classification, nitroglycerin dosage, SAQ questionnaire), exertional capacity (6MWT), quality of life (SF-36 questionnaire) and imaging evaluation (myocardial perfusion imaging and echocardiography). Safety outcome include the change of serum TNT, CKMB, BNP and adverse event (AE) occurrence. The participants will be followed up at 13th week, 6th months and 12th months.

DETAILED DESCRIPTION:
CAD is a challenging affliction which has a high annual morbidity rate in China and the world. Severe CAD may lead to compromised cardiac function, decreased exertional capacity and poor quality of life (QOL). The most common treatment for CAD is medication, percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG). However, some patients had long-term of history with complex severe artery lesions, they are not candidate for redo interventional therapy. Cardiac shock wave therapy (CSWT) is an exploring therapy used globally for CAD patients, which is known for its safety, non-invasiveness and effectiveness. In the previous clinical studies, CSWT can alleviated angina symptom, improved myocardial ischemia and increased exertional capacity. Many single arm studies proved its efficacy and safety. Our RCT has already finished, and results are in submission processing.

This is a prospective, single arm, observational study design. CAD patients will be enrolled consecutively. The entire treatment period will last 3 months with 9 sessions. CSWT will be administered in the first week, follow by a 3-week non-treatment interval. Outcomes are assessed as efficacy outcomes and safety outcomes. Efficacy outcomes include symptom (CCS score, NYHA classification, nitroglycerin dosage, SAQ questionnaire), exertional capacity (6MWT), quality of life (SF-36 questionnaire) and imaging evaluation (myocardial perfusion imaging and echocardiography). Safety outcome include the change of serum TNT, CKMB, BNP and adverse event (AE) occurrence. Symptom, 6MWT and questionnaires will be evaluated at baseline and 13th week, 6th months, 12th months of CSWT. Imaging outcomes will be evaluated at baseline and 13th week, 12th months of CSWT. The level of TNT, CKMB and BNP will be tested before and 1st week after initiation of CSWT.

ELIGIBILITY:
Inclusion Criteria:

* Multiple or diffused coronary artery stenosis via coronary angiography, and not the candidates for PCI or CABG;
* Myocardial ischemia documented by stressed MPI and echocardiography;
* Refractory angina that has not been alleviated after at least three months of optimal medication treatment (OMT);
* Left ventricular ejection fraction (LVEF) ≥ 30%.

Exclusion Criteria:

* Acute myocardial infarction within one month;
* PCI or CABG within one month;
* Heart transplant patient;
* Patients with prosthetic valves;
* Cases of atrial or ventricular thrombosis;
* Uncontrolled heart failure with LVEF <30%;
* Severe arrhythmia; (viii) patients with pacemakers;
* Cases of infective endocarditis;
* Chronic obstructive pulmonary disease patients;
* Pregnant or nursing women;
* Patients with silicone breast implants;
* Chest tumor patients;
* Patients already participating in other clinical trials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe CAD patients were enrolled and coronary angiography indicated complicated severe lesions. Although they were under OMT, stress myocardial perfusion imaging (MPI) showed obvious ischemia. They were not candidate for coronary revascularization.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Summed Rest Score | Change from Baseline Summed Rest Score at 12 months.
  Summed Rest Score of 17 segments of left ventricle under myocardial perfusion imaging. Each segment will be scored from 0 to 4. The minimum score is 0 while the maximum score is 68. Higher score means worse ischemia.
Summed Stress Score | Change from Baseline Summed Stress Score at 12 months.
  Summed Stress Score of 17 segments of left ventricle under myocardial perfusion imaging. Each segment will be scored from 0 to 4. The minimum score is 0 while the maximum score is 51. Higher score means worse ischemia.
Summed Reverse Score | Change from Baseline Summed Reverse Score at 12 months.
  Summed Reverse Score of 17 segments of left ventricle under myocardial perfusion imaging. Each segment will be scored from 0 to 4. The minimum score is 0 while the maximum score is 51. Higher score means worse ischemia.
Regional Rest Score | Change from Baseline Regional Rest Score at 12 months.
  Rest Score of target treatment segments of left ventricle under myocardial perfusion imaging. Each segment will be scored from 0 to 4. The minimum score is 0 while the maximum score is 8. Higher score means worse ischemia.
Regional Stress Score | Change from Baseline Regional Stress Score at 12 months.
  Stress Score of target treatment segments of left ventricle under myocardial perfusion imaging will be calculate. Each segment will be scored from 0 to 4. The minimum score is 0 while the maximum score is 8. Higher score means worse ischemia.
Regional Reverse Score | Change from Baseline Regional Reverse Score at 12 months.
  Reverse Score of target treatment segments of left ventricle under myocardial perfusion imaging will be calculate. Each segment will be scored from 0 to 4. The minimum score is 0 while the maximum score is 8. Higher score means worse ischemia.

SECONDARY OUTCOMES:
CCS score | Change from Baseline CCS score at 12 months.
  Canadian Cardiovascular Society score. The score is from 1 to 4 score. Higher score means worse ischemia.
NYHA classification | Change from Baseline NYHA classification at 12 months.
  Now York Heart Association classification. The score is from 1 to 4. Higher score means worse heart function.
Seattle Angina Questionnaire | Change from Baseline NYHA classification at 12 months.
  Seattle Angina Questionnaire has five domain: physical limitation, angina stability, angina frequency, treatment satisfaction and quality of life. Each domain are 0-100 scale.
QOL: SF-36 Questionnaire | Change from Baseline SF-36 score at 12 months.
  SF-36 Questionnaire include vitality, physical functioning, body pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health. Each items are 0-100 scale.
Six minutes walk test | Change from Baseline 6MWT at 12 months.
  Six minutes walk test proceed according to ATS guideline. The total distance will be recored.
Left ventricular ejection fraction | Change from Baseline status at 12 months
  Left ventricular ejection fraction on echocardiography

OTHER OUTCOMES:
Cardiac enzyme | Change from Baseline status at 13th week after treatment.
  Serum Troponin T, CKMB
Brain Natrium Peptide | Change from Baseline status at 13th week after treatment.
  Serum brain Natrium Peptide

CONTACTS AND LOCATIONS:
Overall Officials: Qing He, MD, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Sorry for that because of policy constraint.

REFERENCES:
- [Result] Zhang Y, Shen T, Liu B, Dai D, Cai J, Zhao C, Du L, Jia N, He Q. Cardiac Shock Wave Therapy Attenuates Cardiomyocyte Apoptosis after Acute Myocardial Infarction in Rats. Cell Physiol Biochem. 2018;49(5):1734-1746. doi: 10.1159/000493616. Epub 2018 Sep 24. PMID 30248666
- [Result] Qiu Q, Shen T, Wang Q, Yu X, Jia N, He Q. Cardiac shock wave therapy protects cardiomyocytes from hypoxia-induced injury by modulating miR-210. Mol Med Rep. 2020 Feb;21(2):631-640. doi: 10.3892/mmr.2019.10892. Epub 2019 Dec 18. PMID 31974607
- [Result] Liu B, Zhang Y, Jia N, Lan M, Du L, Zhao D, He Q. Study of the Safety of Extracorporeal Cardiac Shock Wave Therapy: Observation of the Ultrastructures in Myocardial Cells by Transmission Electron Microscopy. J Cardiovasc Pharmacol Ther. 2018 Jan;23(1):79-88. doi: 10.1177/1074248417725877. Epub 2017 Sep 1. PMID 28862043
- [Result] Du L, Shen T, Liu B, Zhang Y, Zhao C, Jia N, Wang Q, He Q. Shock Wave Therapy Promotes Cardiomyocyte Autophagy and Survival during Hypoxia. Cell Physiol Biochem. 2017;42(2):673-684. doi: 10.1159/000477885. Epub 2017 Jun 15. PMID 28618416
- [Result] Yu W, Shen T, Liu B, Wang S, Li J, Dai D, Cai J, He Q. Cardiac shock wave therapy attenuates H9c2 myoblast apoptosis by activating the AKT signal pathway. Cell Physiol Biochem. 2014;33(5):1293-303. doi: 10.1159/000358697. Epub 2014 Apr 28. PMID 24802592